CLINICAL TRIAL: NCT02726763
Title: Pilot Study of Feasibility and Tolerability of Transcranial Direct Current Stimulation With Concurrent Cognitive Training
Brief Title: Feasibility and Tolerability of Transcranial Direct Current Stimulation With Concurrent Cognitive Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-034
Record Dates: First submitted 2016-03-30; First posted 2016-04-04 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Survivors
Keywords: Transcranial Direct Current Stimulation (tDCS); Cognitive Training; 16-034
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Surveys and Questionnaires

ARMS (1):
- tDCS with cognitive training (Experimental): We will collect: 1) self-reported demographic information (~5 min) 2) cognitive functioning data (PAOFI) at session 1 and session 4 (~10min) [60]; 3) behavioral data and EEG data from the tDCS stimulation task for each session (downloaded by investigators); 4) patient feedback on their experience with tDCS (tDCS Patient Experience Questionnaire (tPEQ)) for each session (~5 min); 5) tDCS accrual and session completion rates at the completion of treatment and 6) Brunoni Adverse Events Questionnaire (~5 min)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Questionnaires

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS)
Behavioral: Questionnaires

SUMMARY:
In this study, the investigators are testing transcranial direct current stimulation (tDCS) in breast cancer survivors. In this pilot study, the investigators want to learn if it is feasible to use this device in memory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors treated with chemotherapy between 40 and 65 years of age with no evidence of disease with treatment completed at least six months prior to study participation with or without current endocrine therapy.
* Self-reported new onset since initiation of treatment cognitive dysfunction as determined by telephone screen using the brief (3 questions) assessment established by Ercoli et al. [3] (endorsement on all three questions):

  1. Do you think or feel that your memory or mental ability has gotten worse since you completed your breast cancer treatment?
  2. Do you think that your mind isn't as sharp now as it was before your breast cancer treatments?
  3. Do you feel like these problems have made it harder to function on your job or take care of things around the home?
* In the judgment of the investigators and/or consenting professional, able to read and comprehend English
* In the judgment of the consenting professional cognitively able to provide informed consent

Exclusion Criteria:

* Patients with prior history of primary Central Nervous System (CNS) cancer or CNS metastases
* As per self report and/or medical record history of diagnosed neurological illness including seizure disorder, a dementing condition, or other neurological illness (multiple sclerosis, history of cerebrovascular accident, etc.)
* Participants with untreated depression or anxiety as assessed by self-report and review of medical history;
* Participants with a history of treated or untreated schizophrenia or bipolar disorder as assessed by self report and review of medical history;
* As per self report participants who are pregnant or who are breastfeeding
* As per self report participants with pacemakers, intracranial electrodes, implanted defibrillators or any other prosthesis.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
number of subjects recruited | 6 months
  feasibility defined by the number of subjects recruited in a six month time frame

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/